CLINICAL TRIAL: NCT02425007
Title: Efficacity of Incentive Spirometry in Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: spiro93
Record Dates: First submitted 2015-04-07; First posted 2015-04-23 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spiro (Experimental): Incentive spirometry
  Interventions: Device: Incentive spirometry
- Control (No Intervention): Control group

INTERVENTIONS:
Device: Incentive spirometry
  Other Names: Coach
  Arms: Spiro

SUMMARY:
The purpose of this study is to evaluate the efficiency of incentive spirometry in elderly. Outcomes are lung function and chest expansion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Pulmonary disease
* Cognitive disorders

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
lung function will be measured by spirometry | 1 month

SECONDARY OUTCOMES:
Chest expansion will be measured by a tape measure | One month

CONTACTS AND LOCATIONS:
Locations (1):
- Brussels, Belgium